CLINICAL TRIAL: NCT01890941
Title: A Late Phase II Study of KCT-0809 in Patients With Dry Eye Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KCT1205
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye syndromes; Corneal diseases; Conjunctival diseases
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases; Conjunctival Diseases

ARMS (3):
- KCT-0809 Lower Dose (Experimental)
  Interventions: Drug: KCT-0809 ophthalmic solution
- KCT-0809 Higher Dose (Experimental)
  Interventions: Drug: KCT-0809 ophthalmic solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KCT-0809 ophthalmic solution
  Arms: KCT-0809 Higher Dose; KCT-0809 Lower Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KCT-0809 compared to placebo in patients with dry eye syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Corneal and conjunctival damage
* Insufficiency of lacrimal secretion
* Ocular symptom

Exclusion Criteria:

* Severe ophthalmic disorder
* Punctual plugs or surgery for occlusion of the lacrimal puncta

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Score of the Corneal conjunctival staining | 8weeks

SECONDARY OUTCOMES:
Incidences of Adverse Events | 8weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo and Other Japanese City, Japan